CLINICAL TRIAL: NCT01737151
Title: Study of 4-Fraction Split-Course Stereotactic Ablative Radiation Therapy of the Treatment of Patients With Low and Intermediate Risk Adenocarcinoma of the Prostate
Brief Title: Stereotactic Body Radiation Therapy in Treating Patients With Low- and Intermediate-Risk Prostate Cancer
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Slow accrual
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MCC-14712; NCI-2012-02545 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2012-11-26; First posted 2012-11-29 (Estimated); Last update posted 2019-09-03 (Actual); Status verified 2019-08

CONDITIONS: Prostate Adenocarcinoma; Stage I Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm I (standard stereotactic body radiation therapy (SBRT) (Active Comparator): Patients undergo standard daily fractions of SBRT over 7-8.5 weeks
  Interventions: Radiation: stereotactic body radiation therapy
- Arm II (four fraction split-course SBRT) (Experimental): Patients undergo 2 fractions of SBRT in weeks 1 and 4
  Interventions: Radiation: four fraction split-course SBRT

INTERVENTIONS:
Radiation: stereotactic body radiation therapy — Undergo SBRT
  Other Names: SBRT, stereotactic radiation therapy, stereotactic radiotherapy
  Arms: Arm I (standard stereotactic body radiation therapy (SBRT)
Radiation: four fraction split-course SBRT — four fraction split-course SBRT
  Arms: Arm II (four fraction split-course SBRT)

SUMMARY:
This clinical trial studies stereotactic body radiation therapy in treating patients with low- and intermediate-risk prostate cancer. Stereotactic body radiation therapy may be able to send x-rays directly to the tumor and cause less damage to normal tissue.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate, in terms of late toxicity, the safety of stereotactic radiation therapy using the proposed fractionation schedule.

SECONDARY OBJECTIVES:

I. To evaluate, in terms of acute toxicity, the safety of stereotactic radiation therapy using the proposed fractionation schedule.

II. To determine stereotactic treatment efficacy through biochemical failure (Phoenix criteria).

III. To determine the protocol completion rate. IV. To describe patient-reported outcomes using International Index of Erectile Function (IIEF) and EPIC Urinary and Bowel Assessment questionnaires.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients undergo standard daily fractions of stereotactic body radiation therapy (SBRT) over 7-8.5 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have low or intermediate risk adenocarcinoma of the prostate as defined by:

  * Low-risk disease - Histopathology score (Gleason sum): =<6, T-stage (per current AJCC staging criteria): T1c-T2a, and PSA: <10
  * Intermediate-risk disease as either:

    * Histopathology score (Gleason sum) =< 6, T-stage (per current American Joint Committee on Cancer [AJCC] staging criteria): T1c-T2a, and prostate-specific antigen (PSA) > 10 but =< 20; or
    * Histopathology score (Gleason sum) 7 with =< 50% of any cores positive, T-stage (per current AJCC staging criteria): T1c-T2a, and PSA < 10
* Charlson index of comorbidity score =< 4
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Patients with history of inflammatory bowel disease, or who require steroid or cytotoxic therapy for collagen vascular disease
* Patients with a history of cancer other than skin cancer within 5 years of the initiation of protocol treatment
* Patients with a history of pelvic irradiation for any reason
* Life expectancy < 10 years - Prior treatment with an anti-androgen, luteinizing hormone-releasing hormone (LHRH) agonist, or a combination of the two
* Prior radiation therapy, brachytherapy, or cryotherapy
* Prior surgical procedure involving peri-rectal and peri-prostatic area

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2013-03-08; Primary Completion 2017-11-09 (Actual); Study Completion 2017-11-09 (Actual)

PRIMARY OUTCOMES:
Late toxicity greater than or equal to grade 2 as defined by the Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 criteria | 2 years
  Will be tested using a continuity corrected chi-square test

SECONDARY OUTCOMES:
Biochemical failure as defined by the Phoenix definition | Up to 5 years
Protocol completion rate | Up to 5 years
  The portion of patients completing the planned protocol with no unacceptable protocol violations is anticipated to be greater than 90%. A completion rate of 70% is deemed unacceptably low.
Patient-reported outcomes | Up to 5 years
  International Index of Erectile Function (IIEF) and Expanded Prostate Cancer Index Composite urinary Assessment (EPIC) urinary and bowel assessments will be used to collect patient-reported outcomes.
  * IIEF is a widely used instrument for the evaluation of male sexual function. It is has been recommended as tool for clinical trials of erectile dysfunction and for diagnostic evaluation of erectile dysfunction severity. 15 questions 1=very low (worst) to 5=very high (best).
  * The EPIC urinary and bowel assessments are comprehensive instruments designed to evaluate urinary and bowel symptoms, thereby providing a unique tool for assessment of quality of life issues important in prostate cancer management. 9 questions 0=no problem to 5=big problem
Acute toxicity greater than or equal to grade 2 as defined by the CTCAE version 4 criteria | Up to 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Timothy J Harris, M.D., Principal Investigator — Massey Cancer Center
Locations (3):
- United States (3):
  - University of Virginia Medical Center, Charlottesville, Virginia
  - Hunter Holmes McGuire VA Medical Center, Richmond, Virginia
  - Virginia Commonwealth University/Massey Cancer Center, Richmond, Virginia